CLINICAL TRIAL: NCT02190188
Title: Effect of Orthotic Devices in the Recovery After Partial Meniscectomy
Brief Title: The Influence of Wedge Insoles After Partial Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Dammerer Dietmar, MD, MD, MSc, PhD, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 602010072014; 602011072014 (Other: Austria:)
Record Dates: First submitted 2014-07-12; First posted 2014-07-15 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Partial Meniscectomy
Keywords: wedge insoles,; knee brace,; orthotic device; goal

ARMS (3):
- No specific treatment (No Intervention): No specific treatment after partial meniscectomy
- Wedge Insole with 5mm wedge angel (Other): Participants wear a wedge insole after partial meniscectomy
  Interventions: Device: Wedge Insole 5mm
- Knee Brace (Other): Participants wear a knee brace after partial meniscectomy
  Interventions: Device: Knee Brace

INTERVENTIONS:
Device: Wedge Insole 5mm
  Arms: Wedge Insole with 5mm wedge angel
Device: Knee Brace
  Arms: Knee Brace

SUMMARY:
Research on the implications of orthotic devices and the recovery after knee arthroscopy are widely known. But only a handful of specific issues have been studied to date. However, the effect of orthotic devices on the recovery after partial meniscectomy are largely unknown. To our best knowledge, there are no studies that deal with the treatment of partial medial or lateral meniscectomy with wedge insoles, valgus or varus knee braces. The purpose of this study is to find out if using wedge inserts or knee orthoses improve the outcomes after partial meniscectomy.

We therefore verify the following hypothesis: In patients with partial meniscectomy can be by the postoperative use of exculpatory wedge deposits or relieving knee brace achieve a significantly better clinical outcome than without specific treatment.

ELIGIBILITY:
Inclusion Criteria:

* full leg x-ray to measure the leg axis
* undersigned Informed Consent Form

Exclusion Criteria:

* at the same time conducted or within one year subsequent corrective osteotomies of the leg axis
* medial meniscectomy combination and valgus
* combination of lateral meniscectomy and varus
* psychiatric or neurological comorbidities that produce a poor compliance
* forth degree cartilage lesions or evident osteoarthritis
* concomitant lesion of the collateral ligaments
* insufficient knowledge of the study language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Knee-specific questionnaires which combine an activity and a quality of life score. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Liebensteiner, Priv. Doz. Mag. Dr. PhD, Principal Investigator — Department of Orthopedic, Medical University of Innsbruck
Locations (1):
- Department of Orthopedic; Medical University of Innsbruck, Innsbruck, Tyrol, Austria